CLINICAL TRIAL: NCT00069537
Title: DirecNet Inpatient Study to Test the Accuracy of Continuous Blood Glucose Monitoring Devices in Children With Type 1 Diabetes
Brief Title: Continuous Glucose Monitors for Children With Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DirecNet 001; HD041890; HD041919-01; HD041908-01; HD041906-01; HD041918-01; HD041915
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes Mellitus, Insulin-Dependent; Type 1 Diabetes; Diabetes in Children; Continuous Glucose Monitoring Devices
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Device: The GlucoWatch® G2™ Biographer (GW2B)
Device: The Continuous Glucose Monitoring System (CGMS™)

SUMMARY:
Good control of blood glucose levels is important in preventing complications from diabetes. This study assessed the accuracy and reliability of two FDA-approved continuous glucose monitors, the Continuous Glucose Monitoring System (CGMS) and the GlucoWatch G2 Biographer (GW2B), in children with type 1 diabetes mellitus (T1DM).

DETAILED DESCRIPTION:
Intensive control of blood glucose levels has been shown to substantially prevent or delay complications of T1DM in adolescents and adults. The major limitation to implementation of intensive glycemic control is hypoglycemia. Younger children may be at increased risk for hypoglycemia and the risk/benefit ratio of intensive glycemic control may be less favorable in this population. Intensive therapy has not been systematically evaluated in children less than 13 years of age. This study was conducted by the Diabetes Research in Children Network (DirecNet) to assess the accuracy of the CGMS and the GW2B glucose monitors in comparison with standard blood glucose measurements in an inpatient setting.

During 24-hour clinical research center stays at five clinical centers, approximately 90 children and adolescents with T1DM (1 to 17 years of age) wore two FDA-approved continuous glucose monitors, CGMS and GW2B, and had frequent serum glucose determinations during the day and night. To assess glucose monitor function during periods of rising and falling blood glucose, insulin-induced hypoglycemia and meal-induced hyperglycemia tests were also performed.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of type 1 diabetes mellitus for at least 1 year prior to study entry
* For children over 2 years of age, body mass index between the 5th and 95th percentile for age and gender
* Weight >= 12 kg (26.5 lbs) if < 7 years of age and >= 16 kg (35 lbs) if >7 years of age
* Normal hematocrit

Exclusion Criteria

* Current use of glucocorticoids
* Skin or other medical disorders that would affect completion of the study
* History of seizures other than those attributable to either hypoglycemia or high fever

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2002-05; Study Completion 2002-11

PRIMARY OUTCOMES:
Accuracy of the GlucoWatch G2 Biographer and CGMS

CONTACTS AND LOCATIONS:
Overall Officials: William V. Tamborlane, MD, Study Chair — Yale University
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Background] Mauras N, Beck R, Ruedy K, Booth A, Weinzimer S, and the Diabetes Research in Children Network (DirecNet) Study Group. The Physiological Variations of Plasma Glucose Concentrations in Healthy, Non-Diabetic Children: Use of Continuous Glucose Sensors. Pediatr Res 2003 Apr;53(4Pt 2):1A-669A
- [Background] Weinzimer S, Beck R, Ruedy K, Booth A, Boland E, and the Diabetes Research in Children Network (DirecNet) Study Group. Mealtime Glycemic Excursions in Pediatric Subjects with Type 1 Diabetes Mellitus (T1DM): The DirecNet Experience.Pediatr Res 2003 Apr;53(4Pt2):1A-669A
- [Background] Tsalikian E, Beck R, Ruedy K, Booth A, Tansey M, and the Diabetes Research in Children Network (DirecNet) Study Group. Glycemic Pattern of Insulin Induced Hypoglycemia in Pediatric Subjects with Type 1 Diabetes Mellitus (T1DM): The DirecNet Experience. Pediatr Res 2003 Apr;53(4Pt2):1A-669A
- [Background] Buckingham B, Beck R, Tamborlane W, Ruedy K, Boland E, Chase P, Wysocki T, Tsalikian E, Wilson D, Mauras N, Weinzimer D, Tansey M, Fiallo-Scharer R, Booth A, Kollman C, and the Diabetes Research In Children Network (DirecNet) Study Group. Diabetes Research in Children Network (DirecNet) Accuracy Study of the Continuous Glucose Monitoring System (CGMS) and GlucoWatch® G2™ Biographer (GWB) in Children with Type 1 Diabetes-A CRC-based Study. Diabetes 2003 Jun;52 Suppl 1:A36.
- [Background] Wilson D, Buckingham B, Beck R, Ruedy K, Kollman C, Tsalikian E, Wysocki T, Weinzimer S, Chase P, and the Diabetes Research in Children Network (DirecNet) Study Group. A 5-center CRC-based Study of the Accuracy of the GlucoWatch®G2™ Biographer in Children and Adolescents with Type 1 Diabetes. Diabetes 2003 Jun;52 Suppl 1:A101.
- [Background] Boland E, Weinzimer S, Beck R, Ruedy K, Kollman C, Buckingham B, Chase P, Tansey M, Mauras N, and the Diabetes Research In Children Network (DirecNet) Study Group. Performance of the Medtronic MiniMed Continuous Glucose Monitoring System (CGMS) in Children with T1DM in the DirecNet Accuracy Study. Diabetes 2003 Jun;52 Suppl 1:A90.
- [Background] Fiallo-Scharer R, Chase P, Beck R, Ruedy K, Booth A, Wysocki T, Boland E, Buckingham B, Tsalikian E, and the Diabetes Research In Children Network (DirecNet) Study Group. Performance of the One Touch Ultra at Different Glucose Levels in Three Age Groups of Children with T1DM in the CRC-DirecNet Accuracy Study. Diabetes 2003 Jun;52 Suppl 1:A562.
- [Background] Diabetes Research in Children Network (DIRECNET) Study Group. The accuracy of the GlucoWatch G2 biographer in children with type 1 diabetes: results of the diabetes research in children network (DirecNet) accuracy study. Diabetes Technol Ther. 2003;5(5):791-800. doi: 10.1089/152091503322526996. PMID 14633344
- [Background] Diabetes Research in Children Network (DIRECNET) Study Group. The accuracy of the CGMS in children with type 1 diabetes: results of the diabetes research in children network (DirecNet) accuracy study. Diabetes Technol Ther. 2003;5(5):781-9. doi: 10.1089/152091503322526987. PMID 14633343
- [Background] Diabetes Research In Children Network (Direcnet) Study Group. A multicenter study of the accuracy of the One Touch Ultra home glucose meter in children with type 1 diabetes. Diabetes Technol Ther. 2003;5(6):933-41. doi: 10.1089/152091503322640971. PMID 14709195
- [Background] Diabetes Research in Children Network (DirecNet) Study Group. Accuracy of the GlucoWatch G2 Biographer and the continuous glucose monitoring system during hypoglycemia: experience of the Diabetes Research in Children Network. Diabetes Care. 2004 Mar;27(3):722-6. doi: 10.2337/diacare.27.3.722. PMID 14988292
- [Background] Tsalikian E, Kollman C, Mauras N, Weinzimer S, Buckingham B, Xing D, Beck R, Ruedy K, Tamborlane W, Fiallo-Scharer R; Diabetes Research in Children Network (DirecNet) Study Group. GlucoWatch G2 Biographer alarm reliability during hypoglycemia in children. Diabetes Technol Ther. 2004 Oct;6(5):559-66. doi: 10.1089/dia.2004.6.559. PMID 15628809
- [Background] Tsalikian E, Beck RW, Kalajian A, Janz KF, Tansey MJ; Diabetes Research in Children Network (DirecNet) Study Group. Function of the GlucoWatch G2 Biographer during exercise. Diabetes Technol Ther. 2005 Feb;7(1):230. doi: 10.1089/dia.2005.7.230. No abstract available. PMID 15738721
- [Background] Buckingham B, Block J, Burdick J, Kalajian A, Kollman C, Choy M, Wilson DM, Chase P; Diabetes Research in Children Network. Response to nocturnal alarms using a real-time glucose sensor. Diabetes Technol Ther. 2005 Jun;7(3):440-7. doi: 10.1089/dia.2005.7.440. PMID 15929675